CLINICAL TRIAL: NCT07109232
Title: Hemodynamic Effects of Surgical Positioning in Patients Undergoing Percutaneous Nephrolithotomy: A Prospective Study
Brief Title: Surgical Position and Hemodynamics in PCNL
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Erkan Cem ÇELİK, Associate Professor MD., Ataturk University
Other Study IDs: Ataunihemo
Record Dates: First submitted 2025-07-22; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Hemodynamic Changes; Surgical Positioning; Percutaneous Nephrolithotomy (PCNL)
Keywords: Nephrolithotomy; Hemodynamics; Surgical position; Monitoring

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemodynamic Response to Position Changes: Hemodynamic variables-including mean arterial pressure (MAP), heart rate (HR), cardiac index (CI), stroke volume index (SVI), pulse pressure variation (PPV), stroke volume variation (SVV), dP/dtmax, arterial elastance (Ea), cardiac cycle efficiency (CCE), and cardiac power index (CPI)-were continuously monitored. Hemodynamic measurements were obtained at six predefined time points using the Pressure Recording Analytical Method (PRAM).
  The first three measurements were recorded during the pre-anesthetic period in the supine, lithotomy, and prone positions, respectively, prior to the induction of anesthesia. The latter three measurements were obtained during the anesthetized period: five minutes after induction while the patient was in the baseline supine position, five minutes after transitioning to the lithotomy position (prior to ureteral catheter placement), and five minutes after repositioning to the prone position, before surgical incision.
  Interventions: Other: Position the patient

INTERVENTIONS:
Other: Position the patient — In addition, prior to the operation and throughout the PCNL procedure, hemodynamic measurements were obtained while patients were positioned in the supine, lithotomy, and prone positions, as necessitated by the surgical protocol.

SUMMARY:
This prospective study aims to evaluate the hemodynamic effects of different surgical positions-supine, lithotomy, and prone-in patients undergoing percutaneous nephrolithotomy (PCNL). Hemodynamic parameters are assessed using the Pressure Recording Analytical Method (PRAM) both while patients are awake and under general anesthesia. The study investigates how positioning-independently and in combination with anesthesia-influences cardiovascular function, including mean arterial pressure (MAP), heart rate (HR), cardiac index (CI), stroke volume index (SVI), pulse pressure variation (PPV), stroke volume variation (SVV), cardiac contractility parameters (dP/dtmax), arterial elastance (Ea), cardiac power index (CPI), and cardiac cycle efficiency (CCE). The findings are expected to contribute to optimizing perioperative management and enhancing patient safety during PCNL procedures.

DETAILED DESCRIPTION:
This prospective clinical trial investigates the hemodynamic effects of different surgical positions-supine, lithotomy, and prone-in patients undergoing percutaneous nephrolithotomy (PCNL). The study evaluates hemodynamic variables both in the awake state and under general anesthesia to distinguish the individual and combined impacts of anesthesia and patient positioning on cardiovascular function.

Hemodynamic measurements are performed using the Pressure Recording Analytical Method (PRAM), a minimally invasive technique that allows continuous assessment of parameters such as mean arterial pressure (MAP), heart rate (HR), cardiac index (CI), pulse pressure variation (PPV), stroke volume variation (SVV), stroke volume index (SVI), cardiac contractility parameters (dP/dtmax), arterial elastance (Ea), cardiac power index (CPI), and cardiac cycle efficiency (CCE). Each patient is sequentially positioned in the three surgical positions while awake, and the same measurements are repeated after the induction of general anesthesia in the corresponding positions.

The primary aim is to determine how surgical positioning under general anesthesia alters key cardiovascular parameters. Secondary objectives include comparing hemodynamic changes across positions in both conscious and anesthetized states, identifying potential risks associated with specific positions, and guiding intraoperative patient management to improve safety and outcomes in PCNL procedures.

The study is conducted at a single center and includes adult patients with ASA physical status I-II scheduled for elective PCNL surgery. The findings are expected to provide valuable data for anesthesiologists and surgeons to optimize perioperative cardiovascular stability, particularly during position changes in urological surgeries.

ELIGIBILITY:
Inclusion Criteria:

Participants must be between 18 and 65 years of age. Participants must have a body mass index (BMI) of less than 30 kg/m². Participants must be classified as American Society of Anesthesiologists (ASA) physical status I or II.

Participants must be scheduled to undergo elective percutaneous nephrolithotomy (PCNL) surgery.

Exclusion Criteria:

Participants with a known history of cardiac disease, including arrhythmia, valvular heart disease, prior cardiac surgery, presence of a pacemaker, or an implanted cardiac defibrillator, will be excluded.

Participants with renal failure will be excluded. Participants who received colloid fluid administration prior to surgery will be excluded.

Participants using vasoactive or inotropic drugs will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18-65 years, classified as ASA physical status I-II, with BMI < 30, undergoing elective percutaneous nephrolithotomy (PCNL) under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Evaluate the effects of supine, lithotomy, and prone position on cardiac cycle efficiency (CCE) during the anesthetic period. | Intraoperative period (under general anesthesia) at three predefined time points: 1) 5 minutes after anesthesia induction in the supine position 2) 5 minutes after transitioning to lithotomy position 3) 5 minutes after repositioning to prone position
  The primary objective was to evaluate the effects of different surgical positions on cardiac cycle efficiency (CCE), a parameter derived from pulse contour analysis during the anesthetic period. First measurement was recorded five minutes after anesthesia induction, while the patient was in the baseline supine position. Second measurement was recorded five minutes after transitioning to the lithotomy position, prior to ureteral catheter insertion. The third measurement was recorded five minutes after repositioning to the prone position

SECONDARY OUTCOMES:
Mean Arterial Pressure assessment | Pre-anesthetic period at three predefined time points: 1) Before anesthesia induction in the supine position 2) 5 minutes after transitioning to lithotomy position (while still awake) 3) 5 minutes after transitioning to prone position (before induction)
  Mean Arterial Pressure (MAP), derived via the PRAM method, was assessed in awake patients at three predefined surgical positions.
Heart Rate (HR) Assessment | Pre-anesthetic period at three predefined time points: 1) Before anesthesia induction in the supine position, 2) 5 minutes after transitioning to lithotomy position (while still awake) 3) 5 minutes after transitioning to prone position (before induction)
  Heart Rate (HR) was recorded using the PRAM method in awake patients at three predefined surgical positions.
Cardiac Index (CI) Assessment | Pre-anesthetic period at three predefined time points: 1) Before anesthesia induction in the supine position, 2) 5 minutes after transitioning to lithotomy position (while still awake) 3) 5 minutes after transitioning to prone position (before induction)
  Cardiac Index (CI) was measured using the PRAM method in awake patients at three predefined surgical positions.
Stroke Volume Index (SVI) Assessment | Pre-anesthetic period at three predefined time points: 1) Before anesthesia induction in the supine position, 2) 5 minutes after transitioning to lithotomy position (while still awake) 3) 5 minutes after transitioning to prone position (before induction)
  Stroke Volume Index (SVI) was assessed via the PRAM method in awake patients at three predefined surgical positions.
dP/dt max Assessment | Pre-anesthetic period at three predefined time points: 1) Before anesthesia induction in the supine position, 2) 5 minutes after transitioning to lithotomy position (while still awake) 3) 5 minutes after transitioning to prone position (before induction)
  dP/dt max, an index of cardiac contractility, was assessed using the PRAM method in awake patients at three predefined surgical positions.
Arterial Elastance (Ea) Assessment | Pre-anesthetic period at three predefined time points: 1) Before anesthesia induction in the supine position, 2) 5 minutes after transitioning to lithotomy position (while still awake) 3) 5 minutes after transitioning to prone position (before induction)
  Arterial Elastance (Ea) was measured using the PRAM method in awake patients at three predefined surgical positions.
Cardiac Cycle Efficiency (CCE) Assessment | Pre-anesthetic period at three predefined time points: 1) Before anesthesia induction in the supine position, 2) 5 minutes after transitioning to lithotomy position (while still awake) 3) 5 minutes after transitioning to prone position (before induction)
  Cardiac Cycle Efficiency (CCE) was derived using the PRAM method in awake patients at three predefined surgical positions.
Cardiac Power Index (CPI) Assessment | Pre-anesthetic period at three predefined time points: 1) before anesthesia induction in the supine position 2) 5 minutes after transitioning to lithotomy position (while still awake) 3) 5 minutes after transitioning to prone position (before induction)
  Cardiac Power Index (CPI) was assessed using the PRAM method in awake patients at three predefined surgical positions.
Mean Arterial Pressure (MAP) Assessment under General Anesthesia | Intraoperative period (under general anesthesia) at three predefined time points: 1) 5 minutes after anesthesia induction in the supine position 2) 5 minutes after transitioning to lithotomy position 3) 5 minutes after repositioning to prone position
  Mean Arterial Pressure (MAP) was measured using the PRAM method in patients under general anesthesia at three surgical positions in the operating room
Heart Rate (HR) Assessment under General Anesthesia | Intraoperative period (under general anesthesia) at three predefined time points: 1) 5 minutes after anesthesia induction in the supine position 2) 5 minutes after transitioning to lithotomy position 3) 5 minutes after repositioning to prone position
  Heart Rate (HR) was recorded using the PRAM method in patients under general anesthesia at three surgical positions in the operating room.
Cardiac Index (CI) Assessment under General Anesthesia | Intraoperative period (under general anesthesia) at three predefined time points: 1) 5 minutes after anesthesia induction in the supine position 2) 5 minutes after transitioning to lithotomy position 3) 5 minutes after repositioning to prone position
  Cardiac Index (CI) was assessed using the PRAM method in patients under general anesthesia at three surgical positions in the operating room.
Stroke Volume Index (SVI) Assessment under General Anesthesia | Intraoperative period (under general anesthesia) at three predefined time points: 1) 5 minutes after anesthesia induction in the supine position 2) 5 minutes after transitioning to lithotomy position 3) 5 minutes after repositioning to prone position
  Stroke Volume Index (SVI) was measured using the PRAM method in patients under general anesthesia at three surgical positions in the operating room.
Pulse Pressure Variation (PPV) Assessment under General Anesthesia | Intraoperative period (under general anesthesia) at three predefined time points: 1) 5 minutes after anesthesia induction in the supine position 2) 5 minutes after transitioning to lithotomy position 3) 5 minutes after repositioning to prone position
  Pulse Pressure Variation (PPV) was measured using the PRAM method in patients under general anesthesia at three surgical positions in the operating room.
Stroke Volume Variation (SVV) Assessment under General Anesthesia | Intraoperative period (under general anesthesia) at three predefined time points: 1) 5 minutes after anesthesia induction in the supine position 2) 5 minutes after transitioning to lithotomy position 3) 5 minutes after repositioning to prone position
  Stroke Volume Variation (SVV) was assessed using the PRAM method in patients under general anesthesia at three surgical positions in the operating room.
dP/dt max Assessment under General Anesthesia | Intraoperative period (under general anesthesia) at three predefined time points: 1) 5 minutes after anesthesia induction in the supine position 2) 5 minutes after transitioning to lithotomy position 3) 5 minutes after repositioning to prone position
  dP/dt max, an index of cardiac contractility, was assessed using the PRAM method in patients under general anesthesia at three surgical positions in the operating room.
Arterial Elastance (Ea) Assessment under General Anesthesia | Intraoperative period (under general anesthesia) at three predefined time points: 1) 5 minutes after anesthesia induction in the supine position 2) 5 minutes after transitioning to lithotomy position 3) 5 minutes after repositioning to prone position
  Arterial Elastance (Ea) was measured using the PRAM method in patients under general anesthesia at three surgical positions in the operating room.
Cardiac Power Index (CPI) Assessment under General Anesthesia | Intraoperative period (under general anesthesia) at three predefined time points: 1) 5 minutes after anesthesia induction in the supine position 2) 5 minutes after transitioning to lithotomy position 3) 5 minutes after repositioning to prone position
  Cardiac Power Index (CPI) was assessed using the PRAM method in patients under general anesthesia at three surgical positions in the operating room.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University Faculty of Medicine, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Background] Lee S, Kim DY, Han J, Kim K, You AH, Kang HY, Park SW, Kim MK, Kim JE, Choi JH. Hemodynamic changes in the prone position according to fluid loading after anaesthesia induction in patients undergoing lumbar spine surgery: a randomized, assessor-blind, prospective study. Ann Med. 2024 Dec;56(1):2356645. doi: 10.1080/07853890.2024.2356645. Epub 2024 May 24. PMID 38794845
- [Background] Romagnoli S, Franchi F, Ricci Z, Scolletta S, Payen D. The Pressure Recording Analytical Method (PRAM): Technical Concepts and Literature Review. J Cardiothorac Vasc Anesth. 2017 Aug;31(4):1460-1470. doi: 10.1053/j.jvca.2016.09.004. Epub 2016 Sep 14. No abstract available. PMID 28012725